CLINICAL TRIAL: NCT06375278
Title: Device to Deliver Intra-Operative Therapeutic Hypothermia for Hearing Preservation in Cochlear Implantation
Brief Title: Investigation of a Device to Deliver Intra-Operative Therapeutic Hypothermia for Hearing Preservation in Cochlear Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restorear Devices LLC (Industry)
Collaborators: University of Miami (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DC019586; 5R44DC019586 (NIH)
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cochlear Implants; Cochlear Implantation; Hearing Loss
Keywords: Cochlear Implant; Residual Hearing; Hearing Preservation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: For the safety study (aim 1), a single group (n=6) will receive the cooling treatment. For the efficacy study (aim 2) patients will be randomized to either a treatment or control arm in a 1:1 ratio (n=24 per group) in a parallel model.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Safety Study (Experimental): Aim 1: Ascertain the safety of the system and device in patients undergoing cochlear implantation (CI). Mild therapeutic hypothermia will be delivered to the subjects during CI surgery via the ear canal.
  Interventions: Device: Intra-Ear Canal Cooling Catheter
- Efficacy Study Cooling (Experimental): Aim 2: Ascertain the applicability and efficacy of the device and system in patients undergoing cochlear implantation (CI). Half of the candidates will receive mild therapeutic hypothermia via the ear canal during cochlear implant surgery.
  Interventions: Device: Intra-Ear Canal Cooling Catheter
- Efficacy Study Control (No Intervention): Aim 2: Ascertain the applicability and efficacy of the device and system in patients undergoing cochlear implantation (CI). Half of the candidates will receive standard of care (no cooling) during cochlear implant surgery.

INTERVENTIONS:
Device: Intra-Ear Canal Cooling Catheter — Mild therapeutic hypothermia will be applied via the catheter device installed inside the ear canal by an experienced surgeon during cochlear implantation (CI) surgery.
  Arms: Efficacy Study Cooling; Safety Study

SUMMARY:
The goal of this interventional clinical study is to investigate the use of mild therapeutic hypothermia for preservation of residual hearing in cochlear implant surgery. The main questions the trial aims to answer are:

1. Is mild therapeutic hypothermia safe for use during cochlear implantation?
2. Is mild therapeutic hypothermia effective at preserving residual hearing after cochlear implantation?

Participants will receive mild therapeutic hypothermia therapy during cochlear implant surgery. Researchers will compare results from those receiving the therapy to those from a control group (individuals receiving no therapy).

DETAILED DESCRIPTION:
Cochlear implants (CI) have dramatically changed the treatment and prognosis for patients with severe to profound sensorineural hearing loss. With the recent advent of electro-acoustic stimulation (EAS), the combined acoustic amplification at low frequencies with electrical stimulation of high frequency cochlear regions promises to benefit patients with even partial residual hearing by improving difficult listening situations like speech-in-noise and music appreciation. Unfortunately, trauma associated with the implant surgery results in inflammation, mechanical and vascular damage, and loss of remaining sensory hair cells (HC) and neurons. As a result, more than 44% of EAS patients lose residual hearing post-CI surgery and the residual hearing deteriorates by more than 30 dB over time in a majority of patients. This loss of residual hearing post-CI surgery has been the primary barrier for an extended application of CI/EAS.

This clinical trial will evaluate a novel mild therapeutic hypothermia device as an effective therapy to preserve residual hearing post-CI. This system does not require modification of the current surgery or CI devices and will deliver localized, controlled mild hypothermia to the sensitive inner ear structures. With preclinical published results, the investigators have already shown that localized hypothermia during CI surgery is highly effective and safe for residual hearing preservation. Here, the investigators will investigate the implementation of a therapy that benefits patients undergoing CI by improving post-surgical audiological outcomes. Extensive prior commercialization and development experience, intellectual property and engineering expertise coupled with the investigators' collaborators' clinical expertise in Otolaryngology and Audiology will ensure the successful clinical and commercial outcome of this therapy.

Overall, the aim of this clinical trial is:

Validate the clinical applicability, safety and efficacy of the system and device assembly for preservation of residual hearing after CI surgery. The device and hypothermia delivery system will be tested on adult patients undergoing CI surgery at the University of Miami. For clinical translation, the investigators aim to demonstrate that the application of hypothermia combined with the current standard of care for cochlear implantation for residual hearing preservation (steroids) is effective. The investigators hypothesize that the hypothermia application will not negatively impact CI function in patients (safety) and will improve early audiologic outcomes (efficacy) compared to the current standard of care in CI surgeries. The investigators will utilize clinically relevant pre-surgical, intra-operative and post-surgical measures in groups of patients receiving the standard of care and hypothermia therapy.

Preliminary and published preclinical data, and an existing system and device have been constructed for this clinical trial. The proposed therapy and device design for CI surgeries represent a non-pharmaceutical therapeutic strategy to preserve residual hearing.

ELIGIBILITY:
Inclusion Criteria:

Potential participants for the study are patients who have been diagnosed with severe to profound hearing loss (HL) and plan to undergo cochlear implantation (CI) at the University of Miami. The cochlear implant surgery, pre and post-surgical care, and activation and programming of the implant are part of the participants' standard of care. If the inclusion criteria are met (age 18 years and older, equal number of men and women, profound sensorineural hearing loss (for safety study n=6) and residual hearing (see criteria below) from pre-surgical auditory brainstem response (ABR) (for efficacy study n=48), equal numbers of CI devices from all 3 manufactures and English or Spanish speakers the patient will be approached by the study personnel and will be asked to participate in the study.

Exclusion Criteria:

Subjects under 18 years of age. Subjects not meeting functional hearing requirements.

Types of CI devices:

The study will enroll patients receiving CI devices from all three manufactures.

1. Advanced Bionics (FDA indications - severe to profound sensorineural hearing loss (greater than or equal to 70 dB HL)

   1. HiRes Ultra 3D slim J
   2. HiRes Ultra 3D midScala
2. Cochlear Corporation (FDA indications - moderate to profound sensorineural hearing loss; sentence recognition less than or equal to 50% in the ear to be implanted AND less than or equal to 60% in the contralateral ear

   1. CI632
   2. CI622
   3. CI612
3. Med-EL (moderately-severe to severe sensorineural hearing loss (greater than or equal to 65 db HL).

   1. Synchrony 2 Flex soft
   2. Synchrony 2 Flex28
   3. Synchrony 2 Flex 24
   4. Synchrony 2 Compressed
   5. Synchrony 2 Medium

Additional patients receiving devices not listed here may be eligible as the criteria by manufacturer change.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pure Tone Audiometry | At initial cochlear implant activation or 1 month post-operatively; 3 and 12 months post-operatively
  Pure-tone average (PTA) of 125, 250 and 500 Hz which will be tested post-operatively in the safety and efficacy arms to measure residual hearing. A clinically significant change in hearing is greater than 10 dB HL (decibels hearing level) shift.

SECONDARY OUTCOMES:
Electrophysiological Impedance | Immediately post-operatively/during surgery; at initial cochlear implant activation/1 month post-operatively; 3 and 12 months post-operatively
  Per standard of care, electrophysiological impedances will be compared between groups intra- and post-operatively to measure CI device and electrode function. Impedances will be measured in the safety and efficacy arms.
Electrically Evoked Compound Action Potential (ECAP) | Immediately post-operatively/during surgery; at initial cochlear implant activation/1 month post-operatively
  Per standard of care, ECAP will be compared between groups intra- and post-operatively to test CI device function. ECAP will be measured in the safety and efficacy arms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lotocki G, de Rivero Vaccari JP, Perez ER, Sanchez-Molano J, Furones-Alonso O, Bramlett HM, Dietrich WD. Alterations in blood-brain barrier permeability to large and small molecules and leukocyte accumulation after traumatic brain injury: effects of post-traumatic hypothermia. J Neurotrauma. 2009 Jul;26(7):1123-34. doi: 10.1089/neu.2008.0802. PMID 19558276
- [Background] Khan AM, Handzel O, Damian D, Eddington DK, Nadol JB Jr. Effect of cochlear implantation on residual spiral ganglion cell count as determined by comparison with the contralateral nonimplanted inner ear in humans. Ann Otol Rhinol Laryngol. 2005 May;114(5):381-5. doi: 10.1177/000348940511400508. PMID 15966525
- [Background] Ye Q, Tillein J, Hartmann R, Gstoettner W, Kiefer J. Application of a corticosteroid (Triamcinolon) protects inner ear function after surgical intervention. Ear Hear. 2007 Jun;28(3):361-9. doi: 10.1097/01.aud.0000261655.30652.62. PMID 17485985
- [Background] Perez E, Viziano A, Al-Zaghal Z, Telischi FF, Sangaletti R, Jiang W, Dietrich WD, King C, Hoffer ME, Rajguru SM. Anatomical Correlates and Surgical Considerations for Localized Therapeutic Hypothermia Application in Cochlear Implantation Surgery. Otol Neurotol. 2019 Oct;40(9):1167-1177. doi: 10.1097/MAO.0000000000002373. PMID 31318786
- [Background] Kurz M, Lyden P, Lundbye J, Rajguru S. Local to Systemic Use of Hypothermia. Ther Hypothermia Temp Manag. 2018 Mar;8(1):4-8. doi: 10.1089/ther.2018.29041.mjk. Epub 2018 Jan 23. No abstract available. PMID 29360005
- [Background] Dugan EA, Bennett C, Tamames I, Dietrich WD, King CS, Prasad A, Rajguru SM. Therapeutic hypothermia reduces cortical inflammation associated with utah array implants. J Neural Eng. 2020 Apr 29;17(2):026035. doi: 10.1088/1741-2552/ab85d2. PMID 32240985
- [Background] Bennett C, Samikkannu M, Mohammed F, Dietrich WD, Rajguru SM, Prasad A. Blood brain barrier (BBB)-disruption in intracortical silicon microelectrode implants. Biomaterials. 2018 May;164:1-10. doi: 10.1016/j.biomaterials.2018.02.036. Epub 2018 Feb 20. PMID 29477707
- [Background] Bennett C, Mohammed F, Alvarez-Ciara A, Nguyen MA, Dietrich WD, Rajguru SM, Streit WJ, Prasad A. Neuroinflammation, oxidative stress, and blood-brain barrier (BBB) disruption in acute Utah electrode array implants and the effect of deferoxamine as an iron chelator on acute foreign body response. Biomaterials. 2019 Jan;188:144-159. doi: 10.1016/j.biomaterials.2018.09.040. Epub 2018 Oct 18. PMID 30343257
- [Background] Tzen YT, Brienza DM, Karg PE, Loughlin PJ. Effectiveness of local cooling for enhancing tissue ischemia tolerance in people with spinal cord injury. J Spinal Cord Med. 2013 Jul;36(4):357-64. doi: 10.1179/2045772312Y.0000000085. PMID 23820151
- [Background] Purdy PD, Novakovic RL, Giles BP, Miller SL, Riegel MS. Spinal cord hypothermia without systemic hypothermia. AJNR Am J Neuroradiol. 2013 Jan;34(1):252-6. doi: 10.3174/ajnr.A3175. Epub 2012 Jul 5. PMID 22766669
- [Background] Dietrich WD, Levi AD, Wang M, Green BA. Hypothermic treatment for acute spinal cord injury. Neurotherapeutics. 2011 Apr;8(2):229-39. doi: 10.1007/s13311-011-0035-3. PMID 21416406
- [Background] Yokobori S, Bullock R, Gajavelli S, Burks S, Mondello S, Mo J, Wang KK, Hayes RL, Bramlett H, Dietrich D. Preoperative-induced mild hypothermia attenuates neuronal damage in a rat subdural hematoma model. Acta Neurochir Suppl. 2013;118:77-81. doi: 10.1007/978-3-7091-1434-6_13. PMID 23564108
- [Background] Matsui T, Ishikawa T, Takeuchi H, Okabayashi K, Maekawa T. Mild hypothermia promotes pro-inflammatory cytokine production in monocytes. J Neurosurg Anesthesiol. 2006 Jul;18(3):189-93. doi: 10.1097/01.ana.0000188639.39844.f6. PMID 16799346
- [Background] Levi AD, Casella G, Green BA, Dietrich WD, Vanni S, Jagid J, Wang MY. Clinical outcomes using modest intravascular hypothermia after acute cervical spinal cord injury. Neurosurgery. 2010 Apr;66(4):670-7. doi: 10.1227/01.NEU.0000367557.77973.5F. PMID 20190669
- [Background] Kawai N, Okauchi M, Morisaki K, Nagao S. Effects of delayed intraischemic and postischemic hypothermia on a focal model of transient cerebral ischemia in rats. Stroke. 2000 Aug;31(8):1982-9; discussion 1989. doi: 10.1161/01.str.31.8.1982. PMID 10926967
- [Background] Dietrich WD, Bramlett HM. The evidence for hypothermia as a neuroprotectant in traumatic brain injury. Neurotherapeutics. 2010 Jan;7(1):43-50. doi: 10.1016/j.nurt.2009.10.015. PMID 20129496
- [Background] Dietrich WD, Atkins CM, Bramlett HM. Protection in animal models of brain and spinal cord injury with mild to moderate hypothermia. J Neurotrauma. 2009 Mar;26(3):301-12. doi: 10.1089/neu.2008.0806. PMID 19245308
- [Background] Deng H, Han HS, Cheng D, Sun GH, Yenari MA. Mild hypothermia inhibits inflammation after experimental stroke and brain inflammation. Stroke. 2003 Oct;34(10):2495-501. doi: 10.1161/01.STR.0000091269.67384.E7. Epub 2003 Sep 11. PMID 12970518
- [Background] Cappuccino A, Bisson LJ, Carpenter B, Marzo J, Dietrich WD 3rd, Cappuccino H. The use of systemic hypothermia for the treatment of an acute cervical spinal cord injury in a professional football player. Spine (Phila Pa 1976). 2010 Jan 15;35(2):E57-62. doi: 10.1097/BRS.0b013e3181b9dc28. PMID 20081503
- [Background] Jiang JY, Lyeth BG, Kapasi MZ, Jenkins LW, Povlishock JT. Moderate hypothermia reduces blood-brain barrier disruption following traumatic brain injury in the rat. Acta Neuropathol. 1992;84(5):495-500. doi: 10.1007/BF00304468. PMID 1462764
- [Background] Lee SM, Zhao H, Maier CM, Steinberg GK. The protective effect of early hypothermia on PTEN phosphorylation correlates with free radical inhibition in rat stroke. J Cereb Blood Flow Metab. 2009 Sep;29(9):1589-600. doi: 10.1038/jcbfm.2009.81. Epub 2009 Jun 24. PMID 19553907
- [Background] Choi JS, Park J, Suk K, Moon C, Park YK, Han HS. Mild Hypothermia Attenuates Intercellular Adhesion Molecule-1 Induction via Activation of Extracellular Signal-Regulated Kinase-1/2 in a Focal Cerebral Ischemia Model. Stroke Res Treat. 2011;2011:846716. doi: 10.4061/2011/846716. Epub 2011 Mar 16. PMID 21716663
- [Background] Fairchild KD, Singh IS, Carter HC, Hester L, Hasday JD. Hypothermia enhances phosphorylation of IkappaB kinase and prolongs nuclear localization of NF-kappaB in lipopolysaccharide-activated macrophages. Am J Physiol Cell Physiol. 2005 Nov;289(5):C1114-21. doi: 10.1152/ajpcell.00152.2005. Epub 2005 Jun 22. PMID 15972840
- [Background] Choi HA, Ko SB, Presciutti M, Fernandez L, Carpenter AM, Lesch C, Gilmore E, Malhotra R, Mayer SA, Lee K, Claassen J, Schmidt JM, Badjatia N. Prevention of shivering during therapeutic temperature modulation: the Columbia anti-shivering protocol. Neurocrit Care. 2011 Jun;14(3):389-94. doi: 10.1007/s12028-010-9474-7. PMID 21210305
- [Background] Lee CH, Van Gelder C, Burns K, Cone DC. Advanced cardiac life support and defibrillation in severe hypothermic cardiac arrest. Prehosp Emerg Care. 2009 Jan-Mar;13(1):85-9. doi: 10.1080/10903120802471907. PMID 19145531
- [Background] Inamasu J, Suga S, Sato S, Horiguchi T, Akaji K, Mayanagi K, Kawase T. Postischemic hypothermia attenuates apoptotic cell death in transient focal ischemia in rats. Acta Neurochir Suppl. 2000;76:525-7. doi: 10.1007/978-3-7091-6346-7_110. PMID 11450083
- [Background] Maier CM, Ahern Kv, Cheng ML, Lee JE, Yenari MA, Steinberg GK. Optimal depth and duration of mild hypothermia in a focal model of transient cerebral ischemia: effects on neurologic outcome, infarct size, apoptosis, and inflammation. Stroke. 1998 Oct;29(10):2171-80. doi: 10.1161/01.str.29.10.2171. PMID 9756600
- [Background] Toyoda T, Suzuki S, Kassell NF, Lee KS. Intraischemic hypothermia attenuates neutrophil infiltration in the rat neocortex after focal ischemia-reperfusion injury. Neurosurgery. 1996 Dec;39(6):1200-5. doi: 10.1097/00006123-199612000-00024. PMID 8938775
- [Background] Wang GJ, Deng HY, Maier CM, Sun GH, Yenari MA. Mild hypothermia reduces ICAM-1 expression, neutrophil infiltration and microglia/monocyte accumulation following experimental stroke. Neuroscience. 2002;114(4):1081-90. doi: 10.1016/s0306-4522(02)00350-0. PMID 12379261
- [Background] Takeda S, Hakuba N, Yoshida T, Fujita K, Hato N, Hata R, Hyodo J, Gyo K. Postischemic mild hypothermia alleviates hearing loss because of transient ischemia. Neuroreport. 2008 Aug 27;19(13):1325-8. doi: 10.1097/WNR.0b013e32830b5f73. PMID 18695517
- [Background] Hyodo J, Hakuba N, Koga K, Watanabe F, Shudou M, Taniguchi M, Gyo K. Hypothermia reduces glutamate efflux in perilymph following transient cochlear ischemia. Neuroreport. 2001 Jul 3;12(9):1983-7. doi: 10.1097/00001756-200107030-00041. PMID 11435934
- [Background] Balkany TJ, Eshraghi AA, Jiao H, Polak M, Mou C, Dietrich DW, Van De Water TR. Mild hypothermia protects auditory function during cochlear implant surgery. Laryngoscope. 2005 Sep;115(9):1543-7. doi: 10.1097/01.mlg.0000173169.45262.ae. PMID 16148692
- [Background] Watanabe F, Koga K, Hakuba N, Gyo K. Hypothermia prevents hearing loss and progressive hair cell loss after transient cochlear ischemia in gerbils. Neuroscience. 2001;102(3):639-45. doi: 10.1016/s0306-4522(00)00510-8. PMID 11226700
- [Background] Henry KR, Chole RA. Hypothermia protects the cochlea from noise damage. Hear Res. 1984 Dec;16(3):225-30. doi: 10.1016/0378-5955(84)90111-4. PMID 6401081
- [Background] Ohlemiller KK, Siegel JH. Cochlear basal and apical differences reflected in the effects of cooling on responses of single auditory nerve fibers. Hear Res. 1994 Nov;80(2):174-90. doi: 10.1016/0378-5955(94)90109-0. PMID 7896576
- [Background] Ohlemiller KK, Siegel JH. The effects of moderate cooling on gross cochlear potentials in the gerbil: basal and apical differences. Hear Res. 1992 Nov;63(1-2):79-89. doi: 10.1016/0378-5955(92)90076-y. PMID 1464578
- [Background] Liberman MC, Dodds LW. Single-neuron labeling and chronic cochlear pathology. II. Stereocilia damage and alterations of spontaneous discharge rates. Hear Res. 1984 Oct;16(1):43-53. doi: 10.1016/0378-5955(84)90024-8. PMID 6511672
- [Background] Brown MC, Smith DI, Nuttall AL. The temperature dependency of neural and hair cell responses evoked by high frequencies. J Acoust Soc Am. 1983 May;73(5):1662-70. doi: 10.1121/1.389387. PMID 6863743
- [Background] Tamames I, King C, Huang CY, Telischi FF, Hoffer ME, Rajguru SM. Theoretical Evaluation and Experimental Validation of Localized Therapeutic Hypothermia Application to Preserve Residual Hearing After Cochlear Implantation. Ear Hear. 2018 Jul/Aug;39(4):712-719. doi: 10.1097/AUD.0000000000000529. PMID 29240567
- [Background] Tamames I, King C, Bas E, Dietrich WD, Telischi F, Rajguru SM. A cool approach to reducing electrode-induced trauma: Localized therapeutic hypothermia conserves residual hearing in cochlear implantation. Hear Res. 2016 Sep;339:32-9. doi: 10.1016/j.heares.2016.05.015. Epub 2016 May 31. PMID 27260269
- [Background] Vivero RJ, Joseph DE, Angeli S, He J, Chen S, Eshraghi AA, Balkany TJ, Van de Water TR. Dexamethasone base conserves hearing from electrode trauma-induced hearing loss. Laryngoscope. 2008 Nov;118(11):2028-35. doi: 10.1097/MLG.0b013e31818173ec. PMID 18818553
- [Background] James DP, Eastwood H, Richardson RT, O'Leary SJ. Effects of round window dexamethasone on residual hearing in a Guinea pig model of cochlear implantation. Audiol Neurootol. 2008;13(2):86-96. doi: 10.1159/000111780. Epub 2007 Nov 29. PMID 18057872
- [Background] Garduno-Anaya MA, Couthino De Toledo H, Hinojosa-Gonzalez R, Pane-Pianese C, Rios-Castaneda LC. Dexamethasone inner ear perfusion by intratympanic injection in unilateral Meniere's disease: a two-year prospective, placebo-controlled, double-blind, randomized trial. Otolaryngol Head Neck Surg. 2005 Aug;133(2):285-94. doi: 10.1016/j.otohns.2005.05.010. PMID 16087029
- [Background] Dinh CT, Chen S, Bas E, Dinh J, Goncalves S, Telischi F, Angeli S, Eshraghi AA, Van De Water T. Dexamethasone Protects Against Apoptotic Cell Death of Cisplatin-exposed Auditory Hair Cells In Vitro. Otol Neurotol. 2015 Sep;36(9):1566-71. doi: 10.1097/MAO.0000000000000849. PMID 26375980
- [Background] Dinh C, Hoang K, Haake S, Chen S, Angeli S, Nong E, Eshraghi AA, Balkany TJ, Van De Water TR. Biopolymer-released dexamethasone prevents tumor necrosis factor alpha-induced loss of auditory hair cells in vitro: implications toward the development of a drug-eluting cochlear implant electrode array. Otol Neurotol. 2008 Oct;29(7):1012-9. doi: 10.1097/MAO.0b013e3181859a1f. PMID 18818545
- [Background] Astolfi L, Guaran V, Marchetti N, Olivetto E, Simoni E, Cavazzini A, Jolly C, Martini A. Cochlear implants and drug delivery: In vitro evaluation of dexamethasone release. J Biomed Mater Res B Appl Biomater. 2014 Feb;102(2):267-73. doi: 10.1002/jbm.b.33004. Epub 2013 Aug 30. PMID 23997036
- [Background] Van De Water TR, Abi Hachem RN, Dinh CT, Bas E, Haake SM, Hoosien G, Vivero R, Chan S, He J, Eshraghi AA, Angeli SI, Telischi FF, Balkany TJ. Conservation of hearing and protection of auditory hair cells against trauma-induced losses by local dexamethasone therapy: molecular and genetic mechanisms. Cochlear Implants Int. 2010 Jun;11 Suppl 1:42-55. doi: 10.1179/146701010X12671178390834. PMID 21756583
- [Background] Eastwood H, Chang A, Kel G, Sly D, Richardson R, O'Leary SJ. Round window delivery of dexamethasone ameliorates local and remote hearing loss produced by cochlear implantation into the second turn of the guinea pig cochlea. Hear Res. 2010 Jun 14;265(1-2):25-9. doi: 10.1016/j.heares.2010.03.006. Epub 2010 Mar 18. PMID 20303400
- [Background] Connolly TM, Eastwood H, Kel G, Lisnichuk H, Richardson R, O'Leary S. Pre-operative intravenous dexamethasone prevents auditory threshold shift in a guinea pig model of cochlear implantation. Audiol Neurootol. 2011;16(3):137-44. doi: 10.1159/000314757. Epub 2010 Jul 29. PMID 20668374
- [Background] Baumgartner WD, Jappel A, Morera C, Gstottner W, Muller J, Kiefer J, Van De Heyning P, Anderson I, Nielsen SB. Outcomes in adults implanted with the FLEXsoft electrode. Acta Otolaryngol. 2007 Jun;127(6):579-86. doi: 10.1080/00016480600987784. PMID 17503226
- [Background] Hochmair I, Hochmair E, Nopp P, Waller M, Jolly C. Deep electrode insertion and sound coding in cochlear implants. Hear Res. 2015 Apr;322:14-23. doi: 10.1016/j.heares.2014.10.006. Epub 2014 Oct 22. PMID 25456089
- [Background] Fitzgerald MB, Sagi E, Jackson M, Shapiro WH, Roland JT Jr, Waltzman SB, Svirsky MA. Reimplantation of hybrid cochlear implant users with a full-length electrode after loss of residual hearing. Otol Neurotol. 2008 Feb;29(2):168-73. doi: 10.1097/mao.0b013e31815c4875. PMID 18165793
- [Background] Dorman MF, Gifford R, Lewis K, McKarns S, Ratigan J, Spahr A, Shallop JK, Driscoll CL, Luetje C, Thedinger BS, Beatty CW, Syms M, Novak M, Barrs D, Cowdrey L, Black J, Loiselle L. Word recognition following implantation of conventional and 10-mm hybrid electrodes. Audiol Neurootol. 2009;14(3):181-9. doi: 10.1159/000171480. Epub 2008 Nov 13. PMID 19005252
- [Background] Yamahara K, Nishimura K, Ogita H, Ito J, Nakagawa T, Furuta I, Kita T, Omori K, Yamamoto N. Hearing preservation at low frequencies by insulin-like growth factor 1 in a guinea pig model of cochlear implantation. Hear Res. 2018 Oct;368:92-108. doi: 10.1016/j.heares.2018.07.004. Epub 2018 Jul 6. PMID 30006113
- [Background] Stathopoulos D, Chambers S, Enke YL, Timbol G, Risi F, Miller C, Cowan R, Newbold C. Development of a safe dexamethasone-eluting electrode array for cochlear implantation. Cochlear Implants Int. 2014 Sep;15(5):254-63. doi: 10.1179/1754762813Y.0000000054. Epub 2014 Jan 3. PMID 24621150
- [Background] Rajan GP, Kuthubutheen J, Hedne N, Krishnaswamy J. The role of preoperative, intratympanic glucocorticoids for hearing preservation in cochlear implantation: a prospective clinical study. Laryngoscope. 2012 Jan;122(1):190-5. doi: 10.1002/lary.22142. PMID 22183635
- [Background] Lyu AR, Kim DH, Lee SH, Shin DS, Shin SA, Park YH. Effects of dexamethasone on intracochlear inflammation and residual hearing after cochleostomy: A comparison of administration routes. PLoS One. 2018 Mar 30;13(3):e0195230. doi: 10.1371/journal.pone.0195230. eCollection 2018. PMID 29601595
- [Background] Haake SM, Dinh CT, Chen S, Eshraghi AA, Van De Water TR. Dexamethasone protects auditory hair cells against TNFalpha-initiated apoptosis via activation of PI3K/Akt and NFkappaB signaling. Hear Res. 2009 Sep;255(1-2):22-32. doi: 10.1016/j.heares.2009.05.003. Epub 2009 May 13. PMID 19442713
- [Background] Green SH, Bailey E, Wang Q, Davis RL. The Trk A, B, C's of neurotrophins in the cochlea. Anat Rec (Hoboken). 2012 Nov;295(11):1877-95. doi: 10.1002/ar.22587. Epub 2012 Oct 8. PMID 23044862
- [Background] Eshraghi AA, Roell J, Shaikh N, Telischi FF, Bauer B, Guardiola M, Bas E, Van De Water T, Rivera I, Mittal J. A novel combination of drug therapy to protect residual hearing post cochlear implant surgery. Acta Otolaryngol. 2016;136(4):420-4. doi: 10.3109/00016489.2015.1134809. Epub 2016 Feb 6. PMID 26854005
- [Background] Eshraghi AA, Adil E, He J, Graves R, Balkany TJ, Van De Water TR. Local dexamethasone therapy conserves hearing in an animal model of electrode insertion trauma-induced hearing loss. Otol Neurotol. 2007 Sep;28(6):842-9. doi: 10.1097/mao.0b013e31805778fc. PMID 17471110
- [Background] Dinh CT, Haake S, Chen S, Hoang K, Nong E, Eshraghi AA, Balkany TJ, Van De Water TR. Dexamethasone protects organ of corti explants against tumor necrosis factor-alpha-induced loss of auditory hair cells and alters the expression levels of apoptosis-related genes. Neuroscience. 2008 Nov 19;157(2):405-13. doi: 10.1016/j.neuroscience.2008.09.012. Epub 2008 Sep 11. PMID 18838114
- [Background] Dinh C, Chen S, Padgett K, Dinh J, Telischi F, Elsayyad N, Johnson P, Angeli S, Bas E, Goncalves S, Eshraghi A, Van De Water T. Dexamethasone Protects Against Radiation-induced Loss of Auditory Hair Cells In Vitro. Otol Neurotol. 2015 Dec;36(10):1741-7. doi: 10.1097/MAO.0000000000000850. PMID 26485588
- [Background] Barkdull GC, Hondarrague Y, Meyer T, Harris JP, Keithley EM. AM-111 reduces hearing loss in a guinea pig model of acute labyrinthitis. Laryngoscope. 2007 Dec;117(12):2174-82. doi: 10.1097/MLG.0b013e3181461f92. PMID 18322422
- [Background] Zou J, Pyykko I, Sutinen P, Toppila E. Vibration induced hearing loss in guinea pig cochlea: expression of TNF-alpha and VEGF. Hear Res. 2005 Apr;202(1-2):13-20. doi: 10.1016/j.heares.2004.10.008. PMID 15811694
- [Background] Radeloff A, Unkelbach MH, Tillein J, Braun S, Helbig S, Gstottner W, Adunka OF. Impact of intrascalar blood on hearing. Laryngoscope. 2007 Jan;117(1):58-62. doi: 10.1097/01.mlg.0000242073.02488.f4. PMID 17202931
- [Background] Pau HW, Just T, Bornitz M, Lasurashvilli N, Zahnert T. Noise exposure of the inner ear during drilling a cochleostomy for cochlear implantation. Laryngoscope. 2007 Mar;117(3):535-40. doi: 10.1097/MLG.0b013e31802f4169. PMID 17334318
- [Background] Jia H, Venail F, Piron JP, Batrel C, Pelliccia P, Artieres F, Uziel A, Mondain M. Effect of surgical technique on electrode impedance after cochlear implantation. Ann Otol Rhinol Laryngol. 2011 Aug;120(8):529-34. doi: 10.1177/000348941112000807. PMID 21922977
- [Background] Havenith S, Lammers MJ, Tange RA, Trabalzini F, della Volpe A, van der Heijden GJ, Grolman W. Hearing preservation surgery: cochleostomy or round window approach? A systematic review. Otol Neurotol. 2013 Jun;34(4):667-74. doi: 10.1097/MAO.0b013e318288643e. PMID 23640087
- [Background] Gstoettner W, Plenk H Jr, Franz P, Hamzavi J, Baumgartner W, Czerny C, Ehrenberger K. Cochlear implant deep electrode insertion: extent of insertional trauma. Acta Otolaryngol. 1997 Mar;117(2):274-7. doi: 10.3109/00016489709117786. PMID 9105465
- [Background] Garcia-Ibanez L, Macias AR, Morera C, Rodriguez MM, Szyfter W, Skarszynski H, Emamdjomeh H, Baumgartner WD. An evaluation of the preservation of residual hearing with the Nucleus Contour Advance electrode. Acta Otolaryngol. 2009 Jun;129(6):651-64. doi: 10.1080/00016480802369278. PMID 18752086
- [Background] Friedland DR, Runge-Samuelson C. Soft cochlear implantation: rationale for the surgical approach. Trends Amplif. 2009 Jun;13(2):124-38. doi: 10.1177/1084713809336422. PMID 19447766
- [Background] Berrettini S, Forli F, Passetti S. Preservation of residual hearing following cochlear implantation: comparison between three surgical techniques. J Laryngol Otol. 2008 Mar;122(3):246-52. doi: 10.1017/S0022215107000254. Epub 2007 Aug 1. PMID 17666134
- [Background] Balkany TJ, Connell SS, Hodges AV, Payne SL, Telischi FF, Eshraghi AA, Angeli SI, Germani R, Messiah S, Arheart KL. Conservation of residual acoustic hearing after cochlear implantation. Otol Neurotol. 2006 Dec;27(8):1083-8. doi: 10.1097/01.mao.0000244355.34577.85. PMID 17130798
- [Background] Bas E, Goncalves S, Adams M, Dinh CT, Bas JM, Van De Water TR, Eshraghi AA. Spiral ganglion cells and macrophages initiate neuro-inflammation and scarring following cochlear implantation. Front Cell Neurosci. 2015 Aug 12;9:303. doi: 10.3389/fncel.2015.00303. eCollection 2015. PMID 26321909
- [Background] O'Leary SJ, Monksfield P, Kel G, Connolly T, Souter MA, Chang A, Marovic P, O'Leary JS, Richardson R, Eastwood H. Relations between cochlear histopathology and hearing loss in experimental cochlear implantation. Hear Res. 2013 Apr;298:27-35. doi: 10.1016/j.heares.2013.01.012. Epub 2013 Feb 5. PMID 23396095
- [Background] Reiss LA, Stark G, Nguyen-Huynh AT, Spear KA, Zhang H, Tanaka C, Li H. Morphological correlates of hearing loss after cochlear implantation and electro-acoustic stimulation in a hearing-impaired Guinea pig model. Hear Res. 2015 Sep;327:163-74. doi: 10.1016/j.heares.2015.06.007. Epub 2015 Jun 16. PMID 26087114
- [Background] Eshraghi AA, Gupta C, Van De Water TR, Bohorquez JE, Garnham C, Bas E, Talamo VM. Molecular mechanisms involved in cochlear implantation trauma and the protection of hearing and auditory sensory cells by inhibition of c-Jun-N-terminal kinase signaling. Laryngoscope. 2013 Mar;123 Suppl 1:S1-14. doi: 10.1002/lary.23902. Epub 2013 Feb 4. PMID 23382052
- [Background] Wanna GB, O'Connell BP, Francis DO, Gifford RH, Hunter JB, Holder JT, Bennett ML, Rivas A, Labadie RF, Haynes DS. Predictive factors for short- and long-term hearing preservation in cochlear implantation with conventional-length electrodes. Laryngoscope. 2018 Feb;128(2):482-489. doi: 10.1002/lary.26714. Epub 2017 Jun 22. PMID 28643327
- [Background] Pfingst BE, Zhou N, Colesa DJ, Watts MM, Strahl SB, Garadat SN, Schvartz-Leyzac KC, Budenz CL, Raphael Y, Zwolan TA. Importance of cochlear health for implant function. Hear Res. 2015 Apr;322:77-88. doi: 10.1016/j.heares.2014.09.009. Epub 2014 Sep 28. PMID 25261772
- [Background] Pfingst BE, Bowling SA, Colesa DJ, Garadat SN, Raphael Y, Shibata SB, Strahl SB, Su GL, Zhou N. Cochlear infrastructure for electrical hearing. Hear Res. 2011 Nov;281(1-2):65-73. doi: 10.1016/j.heares.2011.05.002. Epub 2011 May 14. PMID 21605648
- [Background] O'Connell BP, Hunter JB, Haynes DS, Holder JT, Dedmon MM, Noble JH, Dawant BM, Wanna GB. Insertion depth impacts speech perception and hearing preservation for lateral wall electrodes. Laryngoscope. 2017 Oct;127(10):2352-2357. doi: 10.1002/lary.26467. Epub 2017 Mar 17. PMID 28304096
- [Background] O'Connell BP, Holder JT, Dwyer RT, Gifford RH, Noble JH, Bennett ML, Rivas A, Wanna GB, Haynes DS, Labadie RF. Intra- and Postoperative Electrocochleography May Be Predictive of Final Electrode Position and Postoperative Hearing Preservation. Front Neurosci. 2017 May 29;11:291. doi: 10.3389/fnins.2017.00291. eCollection 2017. PMID 28611574
- [Background] Formeister EJ, McClellan JH, Merwin WH 3rd, Iseli CE, Calloway NH, Teagle HF, Buchman CA, Adunka OF, Fitzpatrick DC. Intraoperative round window electrocochleography and speech perception outcomes in pediatric cochlear implant recipients. Ear Hear. 2015 Mar-Apr;36(2):249-60. doi: 10.1097/AUD.0000000000000106. PMID 25259669
- [Background] Fontenot TE, Giardina CK, Dillon M, Rooth MA, Teagle HF, Park LR, Brown KD, Adunka OF, Buchman CA, Pillsbury HC, Fitzpatrick DC. Residual Cochlear Function in Adults and Children Receiving Cochlear Implants: Correlations With Speech Perception Outcomes. Ear Hear. 2019 May/Jun;40(3):577-591. doi: 10.1097/AUD.0000000000000630. PMID 30169463
- [Background] Nikolopoulos TP, O'Donoghue GM, Archbold S. Age at implantation: its importance in pediatric cochlear implantation. Laryngoscope. 1999 Apr;109(4):595-9. doi: 10.1097/00005537-199904000-00014. PMID 10201747
- [Background] Gantz BJ, Turner CW. Combining acoustic and electrical hearing. Laryngoscope. 2003 Oct;113(10):1726-30. doi: 10.1097/00005537-200310000-00012. PMID 14520097
- [Background] Fitzpatrick DC, Campbell AP, Choudhury B, Dillon MT, Forgues M, Buchman CA, Adunka OF. Round window electrocochleography just before cochlear implantation: relationship to word recognition outcomes in adults. Otol Neurotol. 2014 Jan;35(1):64-71. doi: 10.1097/MAO.0000000000000219. PMID 24317211
- [Background] Carlson ML, Driscoll CL, Gifford RH, Service GJ, Tombers NM, Hughes-Borst BJ, Neff BA, Beatty CW. Implications of minimizing trauma during conventional cochlear implantation. Otol Neurotol. 2011 Aug;32(6):962-8. doi: 10.1097/MAO.0b013e3182204526. PMID 21659922
- [Background] Tobey EA, Thal D, Niparko JK, Eisenberg LS, Quittner AL, Wang NY; CDaCI Investigative Team. Influence of implantation age on school-age language performance in pediatric cochlear implant users. Int J Audiol. 2013 Apr;52(4):219-29. doi: 10.3109/14992027.2012.759666. Epub 2013 Feb 28. PMID 23448124
- [Background] Santa Maria PL, Domville-Lewis C, Sucher CM, Chester-Browne R, Atlas MD. Hearing preservation surgery for cochlear implantation--hearing and quality of life after 2 years. Otol Neurotol. 2013 Apr;34(3):526-31. doi: 10.1097/MAO.0b013e318281e0c9. PMID 23503094
- [Background] Prentiss S, Sykes K, Staecker H. Partial deafness cochlear implantation at the University of Kansas: techniques and outcomes. J Am Acad Audiol. 2010 Mar;21(3):197-203. doi: 10.3766/jaaa.21.3.8. PMID 20211124
- [Background] Kopelovich JC, Reiss LA, Etler CP, Xu L, Bertroche JT, Gantz BJ, Hansen MR. Hearing Loss After Activation of Hearing Preservation Cochlear Implants Might Be Related to Afferent Cochlear Innervation Injury. Otol Neurotol. 2015 Jul;36(6):1035-44. doi: 10.1097/MAO.0000000000000754. PMID 25955750
- [Background] Gantz BJ, Hansen MR, Turner CW, Oleson JJ, Reiss LA, Parkinson AJ. Hybrid 10 clinical trial: preliminary results. Audiol Neurootol. 2009;14 Suppl 1(Suppl 1):32-8. doi: 10.1159/000206493. Epub 2009 Apr 22. PMID 19390173
- [Background] Briggs RJ, Tykocinski M, Saunders E, Hellier W, Dahm M, Pyman B, Clark GM. Surgical implications of perimodiolar cochlear implant electrode design: avoiding intracochlear damage and scala vestibuli insertion. Cochlear Implants Int. 2001 Sep;2(2):135-49. doi: 10.1179/cim.2001.2.2.135. PMID 18792095
- [Background] Ahmad FI, Choudhury B, De Mason CE, Adunka OF, Finley CC, Fitzpatrick DC. Detection of intracochlear damage during cochlear implant electrode insertion using extracochlear measurements in the gerbil. Laryngoscope. 2012 Mar;122(3):636-44. doi: 10.1002/lary.22488. Epub 2012 Jan 17. PMID 22252968
- [Background] Adunka O, Kiefer J, Unkelbach MH, Radeloff A, Gstoettner W. Evaluating cochlear implant trauma to the scala vestibuli. Clin Otolaryngol. 2005 Apr;30(2):121-7. doi: 10.1111/j.1365-2273.2004.00935.x. PMID 15839863
- [Background] Eshraghi AA, Polak M, He J, Telischi FF, Balkany TJ, Van De Water TR. Pattern of hearing loss in a rat model of cochlear implantation trauma. Otol Neurotol. 2005 May;26(3):442-7; discussion 447. doi: 10.1097/01.mao.0000169791.53201.e1. PMID 15891647
- [Background] Bas E, Dinh CT, Garnham C, Polak M, Van de Water TR. Conservation of hearing and protection of hair cells in cochlear implant patients' with residual hearing. Anat Rec (Hoboken). 2012 Nov;295(11):1909-27. doi: 10.1002/ar.22574. Epub 2012 Oct 8. PMID 23044907
- [Background] Wardrop P, Whinney D, Rebscher SJ, Roland JT Jr, Luxford W, Leake PA. A temporal bone study of insertion trauma and intracochlear position of cochlear implant electrodes. I: Comparison of Nucleus banded and Nucleus Contour electrodes. Hear Res. 2005 May;203(1-2):54-67. doi: 10.1016/j.heares.2004.11.006. PMID 15855030
- [Background] Tanaka C, Nguyen-Huynh A, Loera K, Stark G, Reiss L. Factors associated with hearing loss in a normal-hearing guinea pig model of Hybrid cochlear implants. Hear Res. 2014 Oct;316:82-93. doi: 10.1016/j.heares.2014.07.011. Epub 2014 Aug 14. PMID 25128626
- [Background] Wright CG, Roland PS. Vascular trauma during cochlear implantation: a contributor to residual hearing loss? Otol Neurotol. 2013 Apr;34(3):402-7. doi: 10.1097/MAO.0b013e318278509a. PMID 23222961
- [Background] Rebscher SJ, Hetherington A, Bonham B, Wardrop P, Whinney D, Leake PA. Considerations for design of future cochlear implant electrode arrays: electrode array stiffness, size, and depth of insertion. J Rehabil Res Dev. 2008;45(5):731-47. doi: 10.1682/jrrd.2007.08.0119. PMID 18816423
- [Background] Markman TM, Quittner AL, Eisenberg LS, Tobey EA, Thal D, Niparko JK, Wang NY; CDaCI Investigative Team. Language development after cochlear implantation: an epigenetic model. J Neurodev Disord. 2011 Dec;3(4):388-404. doi: 10.1007/s11689-011-9098-z. Epub 2011 Nov 19. PMID 22101809
- [Background] Wanna GB, Noble JH, Carlson ML, Gifford RH, Dietrich MS, Haynes DS, Dawant BM, Labadie RF. Impact of electrode design and surgical approach on scalar location and cochlear implant outcomes. Laryngoscope. 2014 Nov;124 Suppl 6(0 6):S1-7. doi: 10.1002/lary.24728. Epub 2014 May 30. PMID 24764083
- [Background] Hassepass F, Bulla S, Maier W, Laszig R, Arndt S, Beck R, Traser L, Aschendorff A. The new mid-scala electrode array: a radiologic and histologic study in human temporal bones. Otol Neurotol. 2014 Sep;35(8):1415-20. doi: 10.1097/MAO.0000000000000412. PMID 24836594
- [Background] Turner CW, Gantz BJ, Vidal C, Behrens A, Henry BA. Speech recognition in noise for cochlear implant listeners: benefits of residual acoustic hearing. J Acoust Soc Am. 2004 Apr;115(4):1729-35. doi: 10.1121/1.1687425. PMID 15101651
- [Background] Kang SY, Colesa DJ, Swiderski DL, Su GL, Raphael Y, Pfingst BE. Effects of hearing preservation on psychophysical responses to cochlear implant stimulation. J Assoc Res Otolaryngol. 2010 Jun;11(2):245-65. doi: 10.1007/s10162-009-0194-7. Epub 2009 Nov 10. PMID 19902297
- [Background] Gifford RH, Dorman MF, Skarzynski H, Lorens A, Polak M, Driscoll CL, Roland P, Buchman CA. Cochlear implantation with hearing preservation yields significant benefit for speech recognition in complex listening environments. Ear Hear. 2013 Jul-Aug;34(4):413-25. doi: 10.1097/AUD.0b013e31827e8163. PMID 23446225
- [Background] Gfeller KE, Olszewski C, Turner C, Gantz B, Oleson J. Music perception with cochlear implants and residual hearing. Audiol Neurootol. 2006;11 Suppl 1:12-5. doi: 10.1159/000095608. Epub 2006 Oct 6. PMID 17063005
- [Background] Dorman MF, Gifford RH, Spahr AJ, McKarns SA. The benefits of combining acoustic and electric stimulation for the recognition of speech, voice and melodies. Audiol Neurootol. 2008;13(2):105-12. doi: 10.1159/000111782. Epub 2007 Nov 29. PMID 18057874